CLINICAL TRIAL: NCT05546034
Title: Nutrition Screening - Route to a More Practical Method
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Alastair Forbes, Visiting Professor, University of Tartu
Other Study IDs: PKL-127
Record Dates: First submitted 2022-09-08; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Internal Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Standard nutrition screening tools to be compared with routine blood tests — None other than completion of questionnaires one of which would be done in routine practice

SUMMARY:
Observational study. Comparison of existing nutritional screening tools based on questionnaires with blood tests already performed on a routine basis.

No intervention undertaken.

DETAILED DESCRIPTION:
Nutrition screening is of established benefit but is difficult to ensure in ordinary clinical practice. It is relatively labour intensive. The investigation aims to determine whether routinely collected laboratory data could provide comparable information without the need for personnel time. It is known that individual blood tests do not provide sufficient sensitivity or specificity but it is hypothesised that combinations of tests could do so.

Included subjects are those admitted to the University Hospital department of internal medicine. All are eligible other than those subject to protective isolation for infection control (COVID, etc). Data collection is in the form of questionnaires to permit the calculation of 3 tools widely used for screening for malnutrition and malnutrition risk, namely the Malnutrition Universal Screening Tool (MUST), the Nutrition Risk Screening 2002 (NRS-2002) and the Subjective Global Assessment (SGA). Nutritional status is documented by the patient's status according to the international definition provided by the Global Leadership Initiative on Malnutrition (GLIM).

The blood tests already performed on a routine basis are captured to go alongside the nutrition screening tools.

Analysis will aim to determine whether combinations of laboratory data can simulate or replicate the information provided by MUST and NRS2002.

ELIGIBILITY:
Inclusion Criteria:

In-patient in department of internal medicine

Exclusion Criteria:

Unable to complete questionnaire or in protective isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-patient in department of internal medicine
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of new nutrition risk screening tool (devised from 200 patients) by validation in 100 contemporaneous patients in comparison with established screening tools (MUST, NRS-2002 and SGA) and malnutrition defined by GLIM. | Within 6 months of completion of recruitment
  Established tools for screening and assessing nutritional status are utilised. These are the Malnutrition Universal Screening Tool (MUST), the Nutrition Risk Screening-2002 (NRS-2002), the Subjective Global Assessment (SGA) and the Global Leadership Initiative on Malnutrition (GLIM). Data from laboratory testing that has already been performed on these patients is extracted from their hospital records. It is hypothesised that multivariate analysis of indicative parameters will identify 6 to 12 tests that can be combined (with appropriate weighting) into a new predictive score.
  300 sets of patient data will be divided on a randomised basis into a group of 200 from whom the prospective new scoring system will be devised, and a group of 100 in whom the score will be tested for validity against NRS-2002.

SECONDARY OUTCOMES:
Validation of new score against GLIM | Within 6 months of completion of recruitment
  The intended new score will be tested against GLIM. The primary validation is against NRS-2002 as the score is intended as a screening tool for high risk of malnutrition, but it is important to determine whether it is also a test of established malnutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- Tartu Ülikooli Kliinikum, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT05546034/Prot_000.pdf